CLINICAL TRIAL: NCT05177952
Title: The Chronic Effects of Low-Load Blood Flow Restriction or Standard of Care Resistance Exercise on Muscle and Neuromuscular Function in Patients With Multiple Sclerosis
Brief Title: Low-Load Blood Flow Restriction on Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003396: BFR MS
Record Dates: First submitted 2021-12-08; First posted 2022-01-05 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Training Study; Multiple Sclerosis; Blood Flow Restriction
Keywords: Blood Flow Restriction; Multiple Sclerosis; Exercise
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Blood Flow Restriction Therapy; Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized between group parallel
Masking Description: Participants and Investigators will be aware of treatment groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Flow Restriction (Experimental): The BFR group will complete 1 set of 30 (1 x 30) at 30% of their 1 repetition maximum for leg press, leg extension, leg curl, chest press, seated row, and shoulder press completed on exercise machines with 2 minutes between exercises.
  Interventions: Other: Blood Flow Restriction
- Standard of Care (Active Comparator): The standard of care group will complete 1 set of 8-12 repetitions at 60-80% of their 1 repetition maximum for leg press, leg extension, leg curl, chest press, seated row, and shoulder press completed on exercise machines with 2 minutes between exercises.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Blood Flow Restriction — Resistance training with BFR
  Arms: Blood Flow Restriction
Other: Standard of Care — Resistance Training with no BFR
  Arms: Standard of Care

SUMMARY:
This research is being done to compare the current standard of care for strength training for patients with Multiple Sclerosis to lightweight resistance training with blood flow restriction.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effectiveness of the current Multiple Sclerosis standard of care exercise recommendations to low-load resistance training with blood flow restriction on functional outcomes, strength, muscle size, and neuromuscular control in Multiple Sclerosis patients. This study involves completing 2 training sessions per week for 12 weeks as well as pre- and post-training assessment visits for a total of 29 visits over 14 weeks. All visits will be on UCF's campus with a member of the research team.

ELIGIBILITY:
Inclusion Criteria:

* Females between the ages of 18 to 55
* Diagnosed with Multiple Sclerosis
* Expanded Disability Status Score of 0 to 6.5
* Able to walk 10 meters without assistance
* Are willing to come in for all 29 testing visits over 14 weeks

Exclusion Criteria:

* No other known cardiovascular, pulmonary, metabolic, muscular, and/or coronary heart disease
* Multiple Sclerosis relapse in the past 30 days
* Are not currently undergoing a rehabilitation protocol
* Are not currently seeking medical care for a chronic condition that could limit exercise capacity other than multiple sclerosis
* Are not currently pregnant

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 20 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Functional Outcomes- 10meter | Day 2, Week 4 and 8, Day 28
  determined via changes in 10 meter walk test, measured by how fast (in minutes and seconds) someone can walk 10 meters
Change in Functional Outcomes- 6min walk | Day 2, Week 4 and 8, Day 28
  determined via changes in 6 minute walk test, measured by how far (in feet) someone can walk in 6 minutes
Change in Functional Outcomes- CST | Day 2, Week 4 and 8, Day 28
  determined via changes in sit-to-stand test, measured by how quickly someone can stand from a seated position
Change in Functional Outcomes- 30CST | Day 2, Week 4 and 8, Day 28
  determined via changes in 30 second sit-to-stand, measured by how many times someone can stand from a seated position in 30 seconds
Change in Functional Outcomes- MFIS | Day 2, Week 4 and 8, Day 28
  determined via changes in Modified Fatigue Impact Scale Questionnaire, sum score of answers on the questionnaire

SECONDARY OUTCOMES:
Changes in Strength | Day 3, Week 4 and 8, Day 29
  determined via maximal voluntary contractions on the Biodex

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Hill, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No